CLINICAL TRIAL: NCT00744887
Title: Phase I, Open-label, Randomized, 3-way Crossover Trial to Assess the Pharmacokinetics of Darunavir (DRV) Given Once-daily With Different Doses of Ritonavir in Healthy Subjects.
Brief Title: TMC114-TiDP3-C181: Study to Assess the Pharmacokinetics of Darunavir (DRV) With Different Doses of Ritonavir in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR015421
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2010-04

CONDITIONS: HIV; AIDS
Keywords: TMC114-TiDP3-C181; TMC114-C181, health volunteers, Darunavir, ritonavir oral solution
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir

INTERVENTIONS:
Drug: Darunavir

SUMMARY:
The objectives are to determine the effect of different ritonavir doses on darunavir (DRV) oral exposure following once-daily oral dosing of DRV/rtv for 7 days, in order to establish an optimal ritonavir boosting dose for DRV and to evaluate short-term safety and tolerability.

DETAILED DESCRIPTION:
This is a Phase I, open-label, randomized (study drug assigned by chance), 3-way crossover trial in healthy volunteers to assess the pharmacokinetics of darunavir (DRV), co-administered with different doses of ritonavir. The trial population will consist of 18 healthy adult volunteers. During 3 subsequent sessions, each volunteer will receive in a randomized way: Treatments A, B and C. In Treatment A, 800 mg DRV once-daily and 100 mg ritonavir once-daily will be administered. In Treatment B, 800 mg DRV once-daily and 50 mg ritonavir once-daily will be administered. In Treatment C, 800 mg DRV once-daily and 20 mg ritonavir once-daily will be administered. All treatments will be administered for 7 days and intake of DRV and ritonavir will be under fed conditions. DRV will be formulated as a 400 mg tablet; ritonavir will be formulated as an oral solution containing 80mg/mL ritonavir. In each treatment session, full pharmacokinetic profiles of DRV and ritonavir will be determined up to 24 hours after administration on Day 1 and up to 72 hours after administration on Day 7. There will be a washout period of at least 7 days between subsequent treatments. Safety and tolerability will be evaluated continuously throughout the trial. During 3 subsequent sessions, each volunteer will receive in a randomized way Treatments A, B and C. In Treatment A, 800/100 mg DRV/rtv once-daily will be administered. In Treatment B, 800/50 mg DRV/rtv once-daily will be administered. In Treatment C, 800/20 mg DRV/rtv once-daily will be administered. All treatments will be administered for 7 days. DRV will be formulated as a 400 mg tablet; ritonavir will be formulated as an oral solution containing 80mg/mL ritonavir.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, electrocardiogram (ECG), vital signs, and the results of blood biochemistry, blood coagulation and hematology tests and a urinalysis carried out at screening

Exclusion Criteria:

* A positive HIV-1 or HIV-2 test at screening
* Hepatitis A, B, or C infection (confirmed by hepatitis A antibody IgM, hepatitis B surface antigen [with a positive hep B PCR], or hepatitis C virus antibody, respectively) at Screening
* Any history of significant skin disease such as, but not limited to, rash or eruptions, food or drug allergy, dermatitis, eczema, psoriasis, folliculitis, or urticaria
* Use of concomitant medication, including over-the-counter products, herbal preparations and dietary supplements. Concomitant medication must have been discontinued at least 14 days before the first dose of trial medication except for paracetamol (acetaminophen), hormone replacement therapy and hormonal contraceptives
* Participation in an investigational drug trial within 60 days prior to the first intake of trial medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To determine the effect of different ritonavir doses (20, 50, 100 mg ritonavir) in DRV oral exposure following once-daily oral dosing of DRV/rtv for 7 days, in order to establish an optimal ritonavir boosting dose for DRV

SECONDARY OUTCOMES:
To evaluate short-term safety and tolerability of DRV following administration of DRV 800 mg once-daily in the presence of different doses of ritonavir for 7 days in healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- See also: Clinical Study Report Synopsis of TMC114-TiDP3-C181: an open-label, randomized, 3-way crossover trial to assess the pharmacokinetics of darunavir (DRV) given once-daily with different doses of ritonavir in healthy subjects. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1015&filename=CR015421_CSR.pdf